CLINICAL TRIAL: NCT01809314
Title: Non-Interventional Study to Evaluate Treatment of Symptomatic Anemia in Patients With Malignancies Receiving Chemo- and NeoRecormon-Therapy
Brief Title: An Observational Study of Epoetin Beta (NeoRecormon) in Participants With Cancer Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21420
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- NeoRecormon in Symptomatic Anemia: Participants with symptomatic anemia who are receiving epoetin beta (NeoRecormon) according to standard of care and the Summary of Product Characteristics will be observed for 4 months. Treatment must be selected at the discretion of the prescriber prior to enrollment and will not be chosen by the Sponsor in this non-interventional study.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — Treatment will be given according to standard of care and the Summary of Product Characteristics during the study.
  Other Names: NeoRecormon

SUMMARY:
This observational study will evaluate the efficacy and safety of epoetin beta (NeoRecormon) in participants with symptomatic anemia and cancer receiving chemotherapy. Participants receiving NeoRecormon once weekly in accordance with the Summary of Product Characteristics will be followed for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Participants with solid tumors or lymphoproliferative disease
* Participants receiving chemotherapy
* Participants for whom erythropoietin is indicated for pre-study Hb level and observed anemic symptoms: Hb less than (<) 11 g/dL or 6.83 millimoles per liter (mmol/L)
* ECOG performance status of 0, 1, or 2

Exclusion Criteria:

* Resistant hypertension
* Acute chronic bleeding within 3 months prior to study
* Iron deficiency that is unmanageable prior to study
* Hypersensitivity to the active substance or any of the excipients of the product
* Pregnant or breastfeeding women
* Epoetin treatment within 6 months prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with symptomatic anemia due to malignancies will be included.
Sampling Method: Probability Sample
Enrollment: 1167 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Hungary (24):
  - Budapest
  - Debrecen
  - Deszk
  - Dunaújváros
  - Eger
  - Farkasgyepű
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Miskolc
  - Mosdós
  - Nyíregyháza
  - Pécs
  - Salgótarján
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Törökbálint
  - Veszprém
  - Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Groups:
- NeoRecormon in Symptomatic Anemia: Participants with symptomatic anemia who received epoetin beta (NeoRecormon) according to standard of care and the Summary of Product Characteristics were observed for 4 months. Treatment was selected at the discretion of the prescriber prior to enrollment and not chosen by the Sponsor in this non-interventional study.
Period: Overall Study
Arm/Group | NeoRecormon in Symptomatic Anemia
Started | 1167
Completed | 422
Not Completed | 745
Not completed — Withdrawal Prior to Treatment | 1
Not completed — Adverse Event | 6
Not completed — Insufficient Therapeutic Response | 14
Not completed — Lost to Follow-up | 724

BASELINE CHARACTERISTICS:
Population: All Participants Enrolled: All participants who were enrolled into the study regardless of whether treatment was received. Number of participants with available data for age = 1134.
Arm/Group | NeoRecormon in Symptomatic Anemia
Number analyzed (Participants) | 1167
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13.0)
Sex/Gender, Customized [Number; unit: participants]
  Male | 398
  Female | 709
  Unknown | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) Level From Baseline to End of Treatment (EOT)
Description: The change in Hb level from Baseline to the EOT visit at Month 4 was averaged among all participants and expressed in grams per liter (g/L).
Time Frame: Baseline, Month 4
Population: All Participants Enrolled; only those who provided data at all study visits were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: g/L
Arm/Group | NeoRecormon in Symptomatic Anemia
Number analyzed (Participants) | 280
g/L | 14.58 [12.684 to 16.478]
Statistical Analysis 1: Comparison: NeoRecormon in Symptomatic Anemia; The difference between Baseline and Month 4 was analyzed using the Wilcoxon signed-rank test; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test

2. Secondary Outcome: Percentage of Participants by Change in Eastern Cooperative Oncology Group (ECOG) Performance Status From Baseline to EOT
Description: ECOG performance status was determined at Baseline and at the EOT visit at Month 4. The assessment used a 3-point scale, including scores of 0 (fully active/able to carry on all pre-disease activities without restriction), 1 (restricted in physically strenuous activity but ambulatory/able to carry out light or sedentary work), or 2 (ambulatory for more than 50% of waking hours and capable of all self care but unable to carry out any work activities). The traditional 6-point scale was not valid because only participants with a performance status of 0, 1, or 2 were eligible for the study. The percentage of participants by change in ECOG performance status was reported. For example, the percentage of participants with ECOG performance status of 0 at Baseline and 2 at EOT is shown in the table as "Baseline 0, EOT 2". Transition to a lower performance status indicates improved/increased independence.
Time Frame: Baseline, Month 4
Population: All Participants Enrolled; only those who provided data at all study visits were included in the analysis. The "Number of Participants Analyzed" reflects the total combined number of participants who provided data for the endpoint. The number of participants used in the denominator for each calculation (n) was based on the ECOG status at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | NeoRecormon in Symptomatic Anemia
Number analyzed (Participants) | 272
percentage of participants
  Baseline 0, EOT 0 (n=71) | 77.5
  Baseline 0, EOT 1 (n=71) | 19.7
  Baseline 0, EOT 2 (n=71) | 2.8
  Baseline 1, EOT 0 (n=168) | 23.8
  Baseline 1, EOT 1 (n=168) | 67.3
  Baseline 1, EOT 2 (n=168) | 8.9
  Baseline 2, EOT 0 (n=33) | 21.2
  Baseline 2, EOT 1 (n=33) | 48.5
  Baseline 2, EOT 2 (n=33) | 30.3
Statistical Analysis 1: Comparison: NeoRecormon in Symptomatic Anemia; Overall (all categories combined) change from Baseline in ECOG performance status at Month 4 was analyzed using Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.001, Wilcoxon signed-rank test

3. Secondary Outcome: Percentage of Participants Who Required Blood Transfusions During the Study
Description: The percentage of participants who required blood transfusions was reported at each assessment visit and was based on the 1-month period preceding the respective visit.
Time Frame: Baseline to Month 1, Month 1 to 2, Month 2 to 3, Month 3 to 4
Population: All Participants Enrolled. The "Number of Participants Analyzed" reflects the total combined number of participants who provided data for the endpoint. The number of participants who provided data for the analysis at each timepoint (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | NeoRecormon in Symptomatic Anemia
Number analyzed (Participants) | 1073
percentage of participants
  Baseline to Month 1 (n=1073) | 4.1
  Month 1 to 2 (n=853) | 4.1
  Month 2 to 3 (n=650) | 3.8
  Month 3 to 4 (n=281) | 3.9

ADVERSE EVENTS:
Time Frame: From Baseline to Month 4
Description: Analysis Population Description: All Participants Enrolled.
Arm/Group | NeoRecormon in Symptomatic Anemia
Serious Adverse Events (participants affected / at risk) | 7/1167
Other Adverse Events (participants affected / at risk) | 6/1167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NeoRecormon in Symptomatic Anemia (N=1167)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Death (General disorders) | 3
Non-Hodgkin's lymphoman (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NeoRecormon in Symptomatic Anemia (N=1167)
Dyspnoea (Cardiac disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Abdominal cavity drainage (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.